CLINICAL TRIAL: NCT02271802
Title: Effect of a Butyrate Enema on the Systemic Concentration of Short Chain Fatty Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: METC 08-2-006
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: SCFA Metabolism
Keywords: Butyrate; Interorgan metabolism; Short-chain fatty acids; Gut production
MeSH Terms: interventions — Butyric Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Butyrate (Experimental): Enema containing sodium butyrate
  Interventions: Dietary Supplement: Sodium butyrate
- Placebo (Placebo Comparator): Enema containing NaCl
  Interventions: Dietary Supplement: NaCl

INTERVENTIONS:
Dietary Supplement: Sodium butyrate — Patients recieved an enema containing butyrate or a placebo during upper abdominal surgery.
  Arms: Butyrate
Dietary Supplement: NaCl
  Arms: Placebo

SUMMARY:
In this placebo-controlled randomized parallel study the effects of a butyrate enema on plasma short-chain fatty acids (SCFA) concentrations and fluxes from portal drained viscera, liver and the splanchnic area are investigated

DETAILED DESCRIPTION:
Patients undergoing upper abdominal surgery are included. During surgery they receive a butyrate enema or placebo enema. Before and after rectal administration, plasma samples are taken from several veins and arteries to analyse SCFA concentrations and fluxes from portal drained viscera, liver and the splanchnic area.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing open liver resection or pancreaticoduodenectomy

Exclusion Criteria:

* known parenchymal liver disease
* presence of ileostomy or colostomy
* patients with inflammatory bowel disease
* antibiotics, prebiotics or probiotics 2 months prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Plasma SCFAs | 0, 5, 15, 30 min after administration

CONTACTS AND LOCATIONS:
Overall Officials: CHC Dejong, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] van der Beek CM, Bloemen JG, van den Broek MA, Lenaerts K, Venema K, Buurman WA, Dejong CH. Hepatic Uptake of Rectally Administered Butyrate Prevents an Increase in Systemic Butyrate Concentrations in Humans. J Nutr. 2015 Sep;145(9):2019-24. doi: 10.3945/jn.115.211193. Epub 2015 Jul 8. PMID 26156796